CLINICAL TRIAL: NCT03624387
Title: Geriatric Inclusive Art: Effects of Painting Sessions on Older In-patients With Cognitive Decline
Acronym: GIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CODIM-FLP-16-292
Record Dates: First submitted 2017-10-30; First posted 2018-08-10 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Impairment
Keywords: older adults, cognitive impairment, art therapy, hospital
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group( No Painting Sessions) (No Intervention): No Geriatric Inclusive Art session.
- Intervention Group( Painting Session) (Experimental): Painting sessions for participants
  Interventions: Other: Painting Sessions

INTERVENTIONS:
Other: Painting Sessions — During the GIA painting session, each participant will be given a white canvas, four brushes and four different colors of painting.Their only instruction will be to cover the white color of the canvas. At the end of each session, the performance of the participants will be evaluated based on their neuropsychological conditions before and after Geriatric Inclusive Art session.
  Arms: Intervention Group( Painting Session)

SUMMARY:
Geriatric Inclusive Art (GIA) painting activity is a new form of art therapy, which has been adapted for older adults hospitalized in medical wards. GIA painting sessions have been associated with a decrease of in-hospital mortality and length of stay, particularly in patients with cognitive impairment. Preservation of a stable health status as well as functionality in activities of daily living of older inpatients is a primary objective of care management, in order to avoid deconditioning, long hospital stays and related higher costs.

DETAILED DESCRIPTION:
1. The introduction of the problem Preservation of a stable health status as well as functionality in activities of daily living of older inpatients is a primary objective of care management, in order to avoid deconditioning, long hospital stays and related higher costs. Geriatric Inclusive Art (GIA) painting sessions have been associated with a decrease of in-hospital mortality and length of stay, particularly in patients with cognitive impairment. A cycle of Geriatric Inclusive Art (GIA) painting sessions could be a complementary and have a synergistic action with usual care provided to older inpatients.
2. The purpose of the study The overall objective of the study is to examine the effects of Geriatric Inclusive Art (GIA) painting sessions on neuropsychological and health conditions in older inpatients with cognitive impairment (i.e.; from mild to severe dementia) admitted in medical wards of the Division of Geriatrics at the Jewish General Hospital (Montreal, Quebec).
3. The motivation for this approach Patients with dementia in a hospital setting are highly vulnerable. Prospective studies show higher rate of adverse outcomes including mortality, delirium, and longer hospital stays. There are limited pharmacological treatment options for demented patients with many adverse effects and the possibility of worsening the illness. Thus, non-pharmacological approaches have their place in the treatment of these patients: they should always be prioritized and used in combination with medication if needed. Art therapy has been used as a non-pharmacological approach in different categories of patients.
4. The general description of the study The study is a clinical trial, single-centered (Jewish General Hospital, Montreal, Quebec), non-randomized, controlled, superiority trial, open, intent-to-treat, with two parallel arms (intervention and control groups), comparative (comparison of two groups of participants: Intervention group which will have GIA painting sessions and control group will have usual care).

This study has been divided into two consecutive periods (i.e.; feasibility and full periods) in order to increase the possibility to show the effects of GIA painting sessions by measuring the right outcomes with the right tools and no lack of power analysis: The feasibility period will last three-months, which will assess the feasibility of measures of outcomes, estimate the magnitude of changes for the primary outcome of the study and the number of sessions needed for a cycle of GIA painting. The full period will consist of the open non-randomized clinical trial to determine effects of GIA painting sessions. This phase will depend on the findings of the feasibility period.

The population recruited in the study, will be older inpatients admitted in medicals wards of Division of Geriatrics at Jewish General Hospital. Inclusion criteria are the following: age of 65 years and older, cognitive impairment corresponding to a dementia from mild to severe stage, regardless the etiology, admission in medicals ward of Division of Geriatrics at Jewish General hospital, medically stable (i.e.; no acute organ failure) patients.

The population will be separated in two groups: Intervention group: participants who will practice GIA painting session, and Control group: participants who will not practice GIA painting sessions. All participants of this group will be matched on Age (± 3 years), sex, reason for admission and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years and older
* Cognitive impairment corresponding to a dementia from mild to severe stage, regardless the sitology. The cognitive impairment is passed on a previous Mini Mental status Examination score of 26 or less
* Admission in medicals ward od Division of Geriatrics at Jewish General Hospital
* Medically stable patients

Exclusion Criteria:

* Younger than 65 years old
* No cognitive impairment, meaning a previous MMSE score of 27 or higher
* Medically unstable
* Infectious preventive measures
* Bed-bound
* Inability to stay in a sitting position in either a chair or a wheelchair, for a minimum of 30 minutes

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
4-Item Neuropsychological Conditions Measure | One hour of session
  Patient's autonomy, behavior, communication, and duty during Geriatric Inclusive Art session.

SECONDARY OUTCOMES:
Change in patient's health conditions associated with number of falls, new acute organ failure during hospitalization, and the number of medication taken by patient. | Up to 6 months
  The information based on medical chart

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada